CLINICAL TRIAL: NCT00270452
Title: Safety of WT1 and PR1 Peptide Vaccination for Patients With Myeloid Malignancies
Brief Title: Safety of Peptide Vaccination for Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060062; 06-H-0062; NCT00313638 (obsolete NCT alias)
Record Dates: First submitted 2005-12-24; First posted 2005-12-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-02-09

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: Myelodyplastic Syndrome (MDS); Wilm's tumor-1; Proteinase-3; Vaccine Therapy; Acute Myeloid Leukemia; Chronic Myeloid Leukemias; Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

INTERVENTIONS:
Drug: WT1 and PR1 Peptide Vaccine

SUMMARY:
This study will test whether certain patients with myelodysplastic syndrome (MDS), acute myeloid leukemia (AML) or chronic myeloid leukemia (CML) can safely be vaccinated with two peptide vaccines derived from proteins called proteinase 3 (PR1) and Wilm's tumor-1 (WT1). These proteins are produced in large amounts by cells of MDS, AML and CML patients. The peptides are combined with an "adjuvant" called Montanide to make the vaccines, and the vaccines are given with GM-CSF (sargramostim). Both Montanide and sargramostim help the immune system respond to the vaccines. The vaccines then activate the immune system to make specialized cells that search out and kill the MDS, AML and CML cells containing the two proteins.

Patients with MDS, AML or CML who are 18 years of age or older may be eligible for this study. Candidates are screened with a medical history and physical examination, blood tests, chest x-ray, and bone marrow aspirate and biopsy. For the bone marrow biopsy, the area of the hip is anesthetized and a special needle is used to draw marrow from the hipbone.

Participants receive an injection (shot) of each peptide vaccine into deep tissue of the upper arm, upper leg, or the abdomen and two separate shots of sargramostim in the same area as the vaccine shots. Patients' vital signs (heart rate, breathing rate, temperature, blood pressure) are measured before and after they receive the vaccines and they are watched for 2 hours after the shots for possible side effects, such as chills, pain at the injection site, stomach upset, allergic reaction, low blood counts, and infection.

Patients return to the clinic 1, 2, 3 and 4 weeks after receiving the vaccines for a brief physical evaluation and blood tests. A chest x-ray is also done at the 4-week visit. Patients may receive whole blood or platelet transfusions if needed to treat the MDS, growth factors (filgrastim, erythropoietin, or others) if needed, and medications to treat any infections that may develop.

DETAILED DESCRIPTION:
Myeloid malignancies including acute myeloid leukemia and the related disorders myelodysplastic syndrome (MDS) and myeloproliferative diseases represent a wide group of bone marrow stem cell malignancies. Some patients can be cured with chemotherapy or by allogeneic stem cell transplantation. However, a proportion of patients progress following chemotherapy and some relapse after transplantation. Therefore, there is need for studies of investigational agents to improve management of these patients.

The immunological graft-versus-leukemia (GVL) effect seen after allogeneic stem cell transplantation suggests that stimulating the patient's own T cell responses to MDS and leukemia with a vaccine might also retard disease progression and even achieve disease remissions. WT1 and PR1 were identified as target antigens because both antigens are highly expressed by CD34+ stem cells of most patients with myeloid malignancies but not by normal marrow cells. An immunotherapeutic approach to vaccinate against PR1 and WT1 antigens could induce T cell response against MDS and leukemic cells while sparing normal cells and by using a combination of two antigens the risk of disease escape by antigen down regulation should be further diminished.

Therefore, we propose to evaluate a vaccine composed of peptides derived from two proteins over-expressed in MDS and leukemia stem cells - proteinase 3 (PR1) and Wilms tumor-1 (WT1). This protocol, the first in a series of planned research, will evaluate the safety of a single dose of a combination of two peptide vaccines, namely PR1:169-177 and WT-1:126-134 in Montanide adjuvant administered concomitantly with GM-CSF (Sargramostim) in select subjects diagnosed with MDS, AML and CML.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosed with FAB subtypes RA, RARS MDS (Low Risk)

OR

Diagnosed with AML and in complete remission within 5 years of treatment with less than 5 percent marrow blasts

OR

Diagnosed with CML In chronic phase

OR

Diagnosed with MDS, AML or CML and are between 6 months-3 years following allogeneic SCT who fulfill the following criteria:

100 percent donor engraftment,

less than 5 percent blasts in marrow

normal marrow cellularity

HLA-A0201 positive at one allele

Ages 18 - 85 years old

EXCLUSION CRITERIA:

Hypoplastic MDS

Relapsed AML

CML in accelerated phase or blast crisis

Relapsed MDS, AML or CML following hematopoietic stem cell transplantation

Hb less than 9 g/dl, neutrophil count less than 1 times 10(9)/1, and/ or platelet count less than 75 times 10(9)/1

Hypocellular bone marrow

History of Wegener's granulomatosis

Serologic antibody against proteinase-3 (ANCA positive)

Previous allergic reaction to montanide adjuvant

Positive test for HIV

Treatment with systemic corticosteroids within 14 days prior to study entry

Co-morbidity of such severity that it would preclude the subject's ability to tolerate protocol therapy

Predicted survival less than 28 days

Pregnant or breast feeding (All female subjects must have a urine pregnancy test within 1 week prior to vaccine administration)

Enrolled in another drug or vaccine clinical trial during the study period

Inability to comprehend the investigational nature of the study and provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-12-22; Primary Completion 2007-10-26 (Actual); Study Completion 2007-10-26 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of and toxicity assoc. with a single dose of a comb. of PR1:169-177 and WT-1:126-134 peptide (in Montanide adjuvant) vaccination admin. concomitantly with GM-CSF (Sargramostim) in selected patients with myeloid malignancie...

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Kato, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Estey EH. Prognosis and therapy of secondary myelodysplastic syndromes. Haematologica. 1998 Jun;83(6):543-9. PMID 9676028
- [Background] Bennett JM, Catovsky D, Daniel MT, Flandrin G, Galton DA, Gralnick HR, Sultan C. Proposals for the classification of the myelodysplastic syndromes. Br J Haematol. 1982 Jun;51(2):189-99. PMID 6952920
- [Background] Vardiman JW, Harris NL, Brunning RD. The World Health Organization (WHO) classification of the myeloid neoplasms. Blood. 2002 Oct 1;100(7):2292-302. doi: 10.1182/blood-2002-04-1199. PMID 12239137
- [Derived] Rezvani K, Yong AS, Mielke S, Savani BN, Musse L, Superata J, Jafarpour B, Boss C, Barrett AJ. Leukemia-associated antigen-specific T-cell responses following combined PR1 and WT1 peptide vaccination in patients with myeloid malignancies. Blood. 2008 Jan 1;111(1):236-42. doi: 10.1182/blood-2007-08-108241. Epub 2007 Sep 17. PMID 17875804